CLINICAL TRIAL: NCT04146597
Title: Short-term Effects of Active Post-training Slider Neural Mobilization on Hamstring Flexibility in Jiu Jitsu Practitioners: a Quasi-experimental Study
Brief Title: Short-term Effects of Active Post-training Slider Neural Mobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Wagner Rodrigues Martins, Professor, University of Brasilia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Slider NM
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Healthy Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neural mobilization (Experimental): The intervention is always performed after Jiu Jitsu practice and at the training site itself. Neural mobilization consisted of the execution of a sciatic nerve sliding technique in three sets of one minute for each lower limb with an interval of one minute between sets, twice a week, for five consecutive weeks, totaling 10 interventions (Garber et al., 2011). The order of the first lower limb to be submitted to the intervention is not standardized, being at the discretion of the subjects.
  Interventions: Other: Neural mobilization

INTERVENTIONS:
Other: Neural mobilization — Neural mobilization (NM) is a physiotherapy method aimed at restoring the dynamic balance between the relative movement of neural tissues and surrounding mechanical interfaces, and different techniques are used for the treatment of various compression syndromes as well as other pain conditions, such as back and neck pain (Basson et al., 2017; Ellis and Hing, 2008). The main techniques used are neurodynamic sliders and neurodynamic tensioners, with the tensioning techniques being considered the more aggressive approach, in which the increase in nerve length occurs (Silva et al., 2014). The neurodynamic sliders techniques are gentle maneuvers as they involve nerve lengthening at one joint and simultaneous reduction in its length at an adjacent joint in order to produce sliding movements of neural structures relative to adjacent tissues (Efstathiou et al., 2015).

SUMMARY:
Jiu Jitsu is a martial art that consists of various techniques that aim to place the opponent in submission. It is essentially a ground fight that requires large movement variety, among which flexibility is a substantial physical aptitude, required to perform specific positions of attack or defence, especially flexibility of the thoracolumbar spine and hamstrings. The literature reports that abnormal posterior lower limb neurodynamics may influence hamstring extensibility and muscle length, and lead to changes in perception of stretch and pain. The objective of the present study is to evaluate the effect of NM, using sliding techniques of the sciatic nerve, immediately after Jiu Jitsu training, on HM flexibility of Jiu Jitsu practitioners. The hypothesis is that NM sliders applied immediately after training would be as effective as an isolated intervention, as demonstrated in soccer players.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults of regular practitioners of Jiu Jitsu;
* Aged between 18 and 59 years;
* Both sexes.

Exclusion Criteria:

* Straight Leg Raise (SLR) test > 75º;
* Hamstrings injury in the previous three months;
* History of any neurological disorder (such as sensory deficits and irradiated pain) or orthopaedics (such as soft tissue or bone injuries) that affected a lower extremity;
* Positive neural tension test (uni or bilateral);
* Fracture in a lower extremity with surgical treatment history in the previous12 months and with conservative treatment in the previous 6 months;
* Herniated lumbar disc diagnosis.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Passive Knee Extension Test (PKE) | 5 week follow up.
  consisting of passive knee extension with hip and knee stabilized at 90º, with the contralateral limb stabilized at the middle third of the thigh and leg by another researcher, and upper limbs along the trunk. From this position passive extension of the knee was performed by the researcher until the patient communicated the sensation of discomfort without pain in the tested hamstrings. This test shows intra-examiner reliability of 0.99.
Straight leg raise test (SLR): | 5 week follow up.
  consisting of raising the limb through passive hip flexion, keeping the knee extended and the subject in the dorsal decubitus position on the mat with both legs extended and upper limbs along the trunk. The assessment of the hip angle was performed by flexing the hip and maintaining the extension of the knee and ankle free, with the contralateral limb stabilized in the middle third of the thigh and leg by another researcher. It is reported that the SLR has a dual function, besides measuring the flexibility of hamstrings it also accesses the sciatic nerve and can test its mobility (Rolls and George, 2004).

CONTACTS AND LOCATIONS:
Overall Officials: Wagner Martins, Principal Investigator — University of Brasilia
Locations (1):
- University of Brasilia, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castellote-Caballero Y, Valenza MC, Martin-Martin L, Cabrera-Martos I, Puentedura EJ, Fernandez-de-Las-Penas C. Effects of a neurodynamic sliding technique on hamstring flexibility in healthy male soccer players. A pilot study. Phys Ther Sport. 2013 Aug;14(3):156-62. doi: 10.1016/j.ptsp.2012.07.004. Epub 2012 Nov 8. PMID 23142014
- [Result] Andreato LV, Lara FJD, Andrade A, Branco BHM. Physical and Physiological Profiles of Brazilian Jiu-Jitsu Athletes: a Systematic Review. Sports Med Open. 2017 Dec;3(1):9. doi: 10.1186/s40798-016-0069-5. Epub 2017 Feb 13. PMID 28194734